CLINICAL TRIAL: NCT05469932
Title: Quantum Molecular Resonance Effects on Patients With Dry Eye Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Asaf Shemer, Physician in the Ophthalmology Department, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAA
Record Dates: First submitted 2022-03-03; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Dry Eye Syndromes
Keywords: Cornea; Dry Eye; Quantum Molecular Resonance
MeSH Terms: conditions — Dry Eye Syndromes; Corneal Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient does not know wheater they are on treatment or placebo arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Pre-treatment medical examination by an ophthalmologist and self-filled questionnaire.
  Four treatment sessions. Each session includes 20 minutes with the instrument active at power level 4. Post-treatment medical examination by an ophthalmologist and self-filled questionnaire.
  Interventions: Device: Rexon device
- Placebo (Placebo Comparator): Pre-treatment medical examination by an ophthalmologist and self-filled questionnaire.
  Four treatment sessions. Each session includes 20 minutes with the instrument active at power level 0. Post-treatment medical examination by an ophthalmologist and self-filled questionnaire.
  Interventions: Device: Rexon device

INTERVENTIONS:
Device: Rexon device — Rexon device for 20 minutes each session. A total of 4 sessions with one week apart from each other.
  Other Names: Resono Ophthalmic

SUMMARY:
The Rexon Eye device (Resono Ophthalmic Inc, Trieste, Italy) is a new device based on QMR technology. Quantum Molecular Resonance (QMR) is a technique in which low-intensity, high-frequency electric currents are administered to a biological tissue through contact electrodes. The device applies stimulation to the epidermis of closed eyelids up to the lid margin by means of specially designed goggles. Previous studies have shown that it is relatively safe with high patient satisfaction. Preliminary studies have also shown it is effective for accelerating healing in chronic wounds and treating dry eye symptoms.

DETAILED DESCRIPTION:
In this study, the investigators aim to examine the efficacy of the Rexon eye device for the treatment of dry eye signs and symptoms in a randomized double-blind placebo-controlled fashion among a cohort of prospectively recruited patients with dry eye. The control group will receive a similar application of treatment with the device goggles disconnected from the device, effectively receiving no treatment. The treatment will be performed by research assistants following thorough instruction by the manufacturing company representatives and/or provided material. Participants will be actively questioned on any harms or side effects in every meeting.

Outcomes will be assessed based on clinical signs and by validated questionnaires on dry eye symptoms (OSDI).

Informed written consent will be obtained from all participants involved in the study prior to enrollment. The goal of the study is to evaluate the Rexon device as a possible additional treatment option for patients with dry eye or to establish it has no added benefit.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 years
* Patients who are willing and able to consent and adhere to the research plan
* Patients diagnosed with dry eye or patients who are at risk for dry eye

Exclusion Criteria:

* Active infection of the eyelid or periorbital area
* Patients who are pregnant or lactating
* Patients under the age of 18
* Those scheduled for (<30 days) or immediately after (<30 days) ocular surgery (excluding cataract and eyelid surgery)
* Patient who do not adhere to all four treatment sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-14 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) Questionnaire | At baseline (pre-intervention) and up to 4 weeks after treatment ends (after-intervention)
  A validated questionnaire that assess the symptoms of ocular irritation in dry eye disease. and how they affect functioning related to vision. This 12-item questionnaire assesses dry eye symptoms and the effects it has on vision-related function in the past week of the patient's life. The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time." A final score is calculated which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease

SECONDARY OUTCOMES:
Change in Meibomian gland dysfunction Grading | At baseline (pre-intervention) and up to 4 weeks after treatment ends (after-intervention)
  Min = 0. Max =4. Low score: low Meibomian gland dysfunction (normal) High score: Meibomian gland dysfunction (pathology)
Change in Corneal Staining | At baseline (pre-intervention) and up to 4 weeks after treatment ends (after-intervention)
  We measure the amount of fluorescein dots (score 0 for 0 dots, score 1 for 1-5 dots, score 2 for 6-30 dots, score 3 for >30 dots) Additional 1 point for - Patches of confluent staining Additional 1 point for - Staining in the pupillary area Additional 1 point for - One or more filament
  Min = 0. Max =6. Low score: Clear cornea (normal) High score: pathological cornea (pathology)
Change in Tear breakup time | At baseline (pre-intervention) and up to 4 weeks after treatment ends (after-intervention)
  Measures the number of seconds for the fluorescein to break and thus assesses the stability of tear film.
  Min = 0. Max = 20. Low score: Tear film instability (pathology) High score: Normal Tear film stability (normal)
Change in Schirmer with anesthesia | At baseline (pre-intervention) and up to 4 weeks after treatment ends (after-intervention)
  The Schirmer's test evaluates aqueous tear production. It is helpful in the assessment of patients with signs and/or symptoms of dry eye - as it can determine whether surface dryness is due to reduced tear production from the lacrimal glands as opposed to some other cause.
  The Schirmer basal secretion test was performed for each patient in both eyes in the following manner: Topical anesthetic was applied to the eye, and the conjunctival fornix was dried with a cotton tip applicator. After a 2-minute waiting period, the paper strip was folded and placed between the lower eyelid and the globe at the junction between the middle and lateral thirds of the eyelid.
  After 5 minutes, the filter paper is removed and the amount of wetting from the fold is measured (mm) We used the standard (no. 41 Whatman) filter paper.
  Min = 0 mm Max = 30 mm Low score: Low tear secretion (pathology) High score: Normal tear secretion (normal)
Change in Corrected visual acuity | At baseline (pre-intervention) and up to 4 weeks after treatment ends (after-intervention)
  LogMAR scale.
  Min = 0. Max = 1. Low score: Normal visual acuity (normal) High score: Imparied visual acuity (pathology)

CONTACTS AND LOCATIONS:
Locations (1):
- Shamir Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Ferrari G, Colucci A, Barbariga M, Ruggeri A, Rama P. High Frequency Electrotherapy for the Treatment of Meibomian Gland Dysfunction. Cornea. 2019 Nov;38(11):1424-1429. doi: 10.1097/ICO.0000000000002063. PMID 31356415
- [Background] Pedrotti E, Bosello F, Fasolo A, Frigo AC, Marchesoni I, Ruggeri A, Marchini G. Transcutaneous periorbital electrical stimulation in the treatment of dry eye. Br J Ophthalmol. 2017 Jun;101(6):814-819. doi: 10.1136/bjophthalmol-2016-308678. Epub 2016 Sep 22. PMID 27660329
- [Background] Sella S, Adami V, Amati E, Bernardi M, Chieregato K, Gatto P, Menarin M, Pozzato A, Pozzato G, Astori G. In-vitro analysis of Quantum Molecular Resonance effects on human mesenchymal stromal cells. PLoS One. 2018 Jan 2;13(1):e0190082. doi: 10.1371/journal.pone.0190082. eCollection 2018. PMID 29293552
- [Derived] Shemer A, Altarescu A, Nusbaum L, Vardi M, Dubinsky-Pertzov B, Hecht I, Or L, Einan-Lifshitz A, Pras E. Quantum Molecular Resonance Effects on Patients With Dry Eye Disease: A Randomized Controlled Trial. Cornea. 2024 Sep 1;43(9):1144-1149. doi: 10.1097/ICO.0000000000003443. Epub 2023 Dec 28. PMID 38166187
- See also: Related Info — https://www.resono.it/

DOCUMENTS (1):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT05469932/Prot_000.pdf